CLINICAL TRIAL: NCT00474331
Title: Genotype-Phenotype Correlation of Multiple Hereditary Exostoses: Multicentre Project
Brief Title: Gene Mutations and Orthopaedic Symptoms Correlation of Multiple Hereditary Exostoses: Multicentre Project
Status: Suspended | Type: Observational
Why Stopped: Due to unavailability of testing for gene mutation
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Other Study IDs: H04-70223
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Exostoses, Multiple Hereditary
Keywords: DNA sequencing; EXT genes; Hereditary Multiple Exostoses,; also known as Multiple Hereditary Exostoses,; also known as Hereditary Multiple Osteochondromas
MeSH Terms: conditions — Exostoses, Multiple Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigator's goal for this project is to examine the causes of the wide variability of the expression of Hereditary Multiple Exostoses (HME). Previous work completed by our group shows that there exists a correlation between genotype and phenotype such that certain mutations or affected genes cause certain patterns of presentation, symptoms, and signs. The investigators intend to achieve this goal by increasing our study sample size to build upon the results generated from the pilot project of this study, in order to obtain statistical significance. This will be achieved by performing genotype-phenotype analysis on new families presenting with HME in British Columbia.

DETAILED DESCRIPTION:
Subject Recruitment:

New patients presenting with HME will be identified through the offices and clinics of British Columbia Children's Hospital Orthopaedic Department. All potential participants will be educated about the study's rationale, purpose, and procedures and informed consent will be obtained.

Demographics:

All probands (affected patient), their first degree family members and extended family members willing to participate in the study will be interviewed. Information including age, gender, ethnic origin, family history, symptoms, complications and previous surgery will be elucidated.

Phenotype:

Affected patients will have their osteochondroma(s) mapped for location, size, morphology, and symptoms. A total of seventy-five phenotypic parameters divided into four major data categories will be collected. The first two categories are accumulated from physical examinations and include stature and limb segment lengths (15 (x2 for left and right). The other two categories, lesion quality (19 parameters) and limb alignment and deformity (26 parameters) will be drawn from radiographic examinations which are part of the patient's current care. All available xrays will be reviewed and the exostoses characterized radiographically. This will establish the patient's genotype.

Genotype:

Each participant whose genotype is unknown will have a 10 cc. blood sample collected at BC Children's Hospital. This sample will be processed for mutation analysis (DNA extraction from blood samples, mutation analysis) at the Clinical Molecular Diagnostic Laboratory at BC Children's Hospital. The techniques used in the pilot study will be implemented with the exception that microsatellite markers will not be used in order to save cost.

Using EXT 1 and EXT 2 primers (Appendix 1) both strands of a DNA segment are sequenced using ABI Big Dye chemistry Version 2. The resulting sequencing reaction products are then run on an ABI 3100 Avant genetic analyzer. Once a sequence is obtained it is analyzed with SeqScape version 2 software which allows comparison with reference sequence.

Data Analysis:

All information resulting from this research study will be kept strictly confidential. All documents will be identified by an ID number and kept in locked filing cabinets. Participants will not be identified by name in any reports of the completed study. Databases will be stored on project-dedicated laptop computer which is locked in the research office.

The phenotypic data collected will be used to describe family degrees (designed using Cyrillic software), phenotypes of affected individuals and mutations in the exostoses genes of interest (site and type of mutation). Subject heights and segment lengths will be converted to percentile figures to standardize for age and gender to allow for comparison amongst groups.

Genotypic data from the mutation analysis of blood samples will include location of the mutation (early in the gene versus late in the gene), type of mutation (alteration of gene as missense, frameshift, nonsense or splice site), and the amino acid change that was caused by the mutation. The data will be analyzed as follows:

Preliminary Analysis

1. EXT 1 versus EXT 2
2. Males versus Females
3. EXT 1 males versus EXT 1 females versus EXT 2 males versus EXT 2 females

   Secondary Analysis
4. Types of mutations (Missense versus Nonsense versus Splice site versus Frameshift)
5. Early or late mutation (less than 1700 base pairs versus greater than 1700 base pairs)

With 2-way analyses, an unpaired t-test will be calculated and with greater than 2-way analyses, an ANOVA will be calculated. Power will be calculated for every comparison due to the huge variation in sample size. Statistical significance will be set to prior at 0.05 and power of 0.8.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HME

Exclusion Criteria

* Subjects residing outside British Columbia for whom genetic testing and X-ray measurements cannot be taken onsite at BC Children's hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New patients presenting with HME will be identified through the offices and clinics of British Columbia Children's Hospital Orthopaedic Department.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2004-06; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
orthopedic symptoms as assessed by X-ray measurements | Post gene mutation identification

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada